CLINICAL TRIAL: NCT03742596
Title: Effect of Probiotics Supplementation on the Side Effects of Radiation Therapy on the Immune System Among Colorectal Cancer Patients
Brief Title: Effect of Probiotics Supplementation on the Side Effects of Radiation Therapy Among Colorectal Cancer Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study was closed without recruitment
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Fawzi Abuhijla, Consultant Radiation Oncologist, King Hussein Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19 KHCC 111
Record Dates: First submitted 2018-11-11; First posted 2018-11-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Radiotherapy; immune system; Inflammatory markers; Life quality
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probiotic Formula Capsule (Experimental): In this intervention arm the patients will receive oral viable capsules of probiotic contain (1*10 10 colony forming unit (CFU)/g) of lactobacillus (Lactobacillus rhamnosus , Lactobacillus acidophilus , Lactobacillus reuteri, Lactobacillus paracasei, Lactobacillus casei, Lactobacillus gasseri, Lactobacillus plantarum) and bifidobacteria (Bifidobacterium lactis, Bifidobacterium breve, Bifidobacterium bifidum, Bifidobacterium longum, Bifidobacterium infantis) species three times a per day
  Interventions: Dietary Supplement: Probiotic Formula Capsule
- Control (Other): In this intervention arm, the control arm will receive normal treatment without any probiotic
  Interventions: Drug: Control

INTERVENTIONS:
Dietary Supplement: Probiotic Formula Capsule — The Probiotic will be coded in a specific label by a researcher. The patient will receive 2 bottles of the drug every 2 weeks and will be followed weekly for 7 weeks.
  Other Names: Treatment
  Arms: Probiotic Formula Capsule
Drug: Control — The Placebos will be coded in a specific label by a researcher.
  Arms: Control

SUMMARY:
Colorectal cancer (CRC) is one of the most common types of cancer worldwide in general and in Jordan in specific. The studies that investigate the role of Probiotics supplementation in improving the inflammatory response, gastrointestinal toxicity and life quality of patients with colorectal cancer during radiotherapy are limited. So, this study aimed to study the effect of probiotics on the response of inflammatory markers, gastrointestinal toxicity, and quality of life in patients with colorectal cancer during radiation therapy.

An interventional double-blind randomized clinical trial (RCT) design will be used in this study. Forty patients will be recruited and assigned either to receive 3 times a day probiotic supplement or to be control with no intervention. The demographic data, anthropometric measurements, Cancer Quality of Life Questionnaire and blood samples will be collected at baseline and at end of radiation therapy. Interleukin-6, interleukin-1,interleukin-10 IL-10, C-reactive protein, tumor necrosis factor-alpha and complete blood count (CBC) will be measured.

The results will approve or disapprove the beneficial effect of using probiotics as adjuvant therapy for CRC patients and other types of cancer to reduce the side effects of radiotherapy and raise body weight as well as improving their quality of life.

DETAILED DESCRIPTION:
To meet the objectives of the study, a control group will be included in parallel with the treatment group in this trail. Forty patients (aged 35-65 years) who recently diagnosed with CRC will be recruited conveniently from the radiation oncology clinic at the King Hussein Cancer Center (KHCC), Amman, Jordan. Patients who meet the inclusion criteria and agree to participate and to take the drug will be allocated to the probiotic supplementation group, while patients who agree to participate but not to receive the drug will be allocated to the control group. The duration of the intervention will be 5 weeks, from the day of radiation until the end of treatment.

For the participants, the King Hussein Cancer Center (KHCC) hospital setting will be utilized for data collection. The patients will be recruited over 12 months and all patients will be asked to sign a written informed consent before enrollment. The patients that will be assigned to the probiotics group (n=20), to receive 3 times a day probiotic supplement. The duration of the intervention (administration of probiotics) will start 10-14 days before radiotherapy and continue over the 5 weeks duration of treatment under the supervision of the treating physician and end with the end of radiation therapy. The blood sample will be collected at baseline and at the end of radiation therapy and 10-14 days after radiation therapy.

The demographic data of each subject will be collected such as; gender, age, body mass index (BMI), tumor location, malignant tumors stage, tumor differentiation, educational level, occupation, family history, smoking, dietary and physical activity. At baseline and end line of the radiation therapy, a Cancer Quality of Life Questionnaire C30 (QLQ-C30) will be collected and blood sample tests will be withdrawn and the following biochemical variables will be measured: immunoglobulin G, immunoglobulin M, immunoglobulin A, interleukin-6 (IL-6), C-reactive protein (CRP), interleukin-1(IL-1), interleukin-10(IL-10), interleukin-12 (IL-12), Tumor necrosis factor-alpha (TNF-α) and complete blood count (CBC).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women,
2. Aged from 35- 65 years with histologically proven CRC and
3. Histologically proven CRC with stage I, II, III
4. Will exposed newly to radiotherapy with the absence of any psychological, sociological or geographical condition that potentially affects the compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

1. Active infection treated by antibiotic therapy or recent infection or recent antibiotic use;
2. Severe cardiovascular and cerebrovascular diseases that could not tolerate radical surgery;
3. Recent use of probiotics, prebiotics, or synbiotic;
4. Evidence of immunodeficiency;
5. Cancer stage IV
6. Pregnancy,
7. Recent/concurrent admission to ER
8. Co-existence of other malignant neoplasms, no other type of cancer in the past 5 years, any serious concomitant systemic disorders or diseases incompatible with the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The level of Immunoglobulin (Ig) A | Through study completion, an average of 1 year
  The level of Immunoglobulin (Ig) A in g/L at both baseline and end line of intervention
The level of Immunoglobulin (Ig) G | Through study completion, an average of 1 year
  The level of Immunoglobulin (Ig) G in g/L at both baseline and end line of intervention
The level of Immunoglobulin (Ig) M | Through study completion, an average of 1 year
  The level of Immunoglobulin (Ig) M in g/L at both baseline and end line of intervention
The Level of Interleukin (IL)-6 | Through study completion, an average of 1 year
  The Level of Interleukin (IL)-6 in pg/ml at both baseline and end line of intervention
The Level of Interleukin (IL)-1 | Through study completion, an average of 1 year
  The Level of Interleukin (IL)-1 in pg/ml at both baseline and end line of intervention
The Level of Interleukin (IL)-10 | Through study completion, an average of 1 year
  The Level of Interleukin (IL)-10 in pg/ml at both baseline and end line of intervention
The Level of Tumor Necrosis Factor (TNF)-α | Through study completion, an average of 1 year
  The Level of TNF-α in pg/ml at both baseline and end line of intervention
The Level of C-reactive protein (CRP) | Through study completion, an average of 1 yea
  The Level of CRP in mg/ml at both baseline and end line of intervention

SECONDARY OUTCOMES:
Quality of Life of patients | Through study completion, an average of 1 year
  The average score of the general quality of life (QoL) subscales assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC-QLQ) which use five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting) range from"Not at A Quite Very" to "Very Much " , and a single global health status/QoL scale range from one (very poor) to 7(Excellent) . In addition, the questionnaire contains five symptom scales that are commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and the perceived financial impact of the disease scale that range from"Not at A Quite Very" to "Very Much ".
The gastrointestinal toxicity | Through study completion, an average of 1 year
  Number and percent of participants with treatment-related adverse events as assessed by NCI Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE) change from baseline in the occurrences and grad of Adverse Events on grading scale at 5 Weeks

OTHER OUTCOMES:
The level of White blood cell count (WBC) | Through study completion, an average of 1 yea
  he level of WBC as cells/ul at both baseline and end line of intervention
The level of red blood cell count (RBC) | Through study completion, an average of 1 yea
  The level of RBC as cells/ul at both baseline and end line of intervention
The mean corpuscular volume (MCV) | Through study completion, an average of 1 yea
  The MCV in fl at both baseline and end line of intervention
The mean corpuscular hemoglobin (MCH) | Through study completion, an average of 1 yea
  The MCH in pg at both baseline and end line of intervention
The mean corpuscular hemoglobin concentration (MCHC) | Through study completion, an average of 1 yea
  The MCH in g/dl at both baseline and end line of intervention
The Platelet count | Through study completion, an average of 1 yea
  The Platelet count as cells/ ul at both baseline and end line of intervention
The of Hemoglobin | Through study completion, an average of 1 yea
  The Hemoglobin in g/dl at both baseline and end line of intervention
The mean platelet volume (MPV) | Through study completion, an average of 1 yea
  The MPV in fl at both baseline and end line of intervention
The level of lymphocytes | Through study completion, an average of 1 yea
  The number of lymphocytes cells at both baseline and end line of intervention
The level of Monocytes | Through study completion, an average of 1 yea
  The number of Monocytes cells at both baseline and end line of intervention
The level of eosinophils | Through study completion, an average of 1 yea
  The number of eosinophils cells at both baseline and end line of intervention
The level of basophils | Through study completion, an average of 1 yea
  The number of basophils cells at both baseline and end line of intervention
The level of neutrophils | Through study completion, an average of 1 yea
  The number of neutrophils cells at both baseline and end line of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi Abuhijla, MD,MSc, Principal Investigator — King Hussein Cancer Center; Lana M Agraib, PhD, Principal Investigator — University of Jordan
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The center (KHCC) where the study conducted emphasis of maintaining privacy and confidentiality of the participants' data

REFERENCES:
- [Background] Abayomi J, Kirwan J, Hackett A. The prevalence of chronic radiation enteritis following radiotherapy for cervical or endometrial cancer and its impact on quality of life. Eur J Oncol Nurs. 2009 Sep;13(4):262-7. doi: 10.1016/j.ejon.2009.02.007. Epub 2009 Jul 28. PMID 19640788
- [Background] Abdollahi H. Probiotic-based protection of normal tissues during radiotherapy. Nutrition. 2014 Apr;30(4):495-6. doi: 10.1016/j.nut.2013.09.006. No abstract available. PMID 24607309
- [Background] Abdollahi, H., Shiri, I., Atashzar, M., Sarebani, M., Moloudi, K., and Samadian, H. (2015), Radiation protection and secondary cancer prevention using biological radioprotectors in radiotherapy. International Journal of Cancer Therapy and Oncology, 3(3).
- [Background] Ambalam P, Raman M, Purama RK, Doble M. Probiotics, prebiotics and colorectal cancer prevention. Best Pract Res Clin Gastroenterol. 2016 Feb;30(1):119-31. doi: 10.1016/j.bpg.2016.02.009. Epub 2016 Feb 19. PMID 27048903
- [Background] Bowen JM, Stringer AM, Gibson RJ, Yeoh AS, Hannam S, Keefe DM. VSL#3 probiotic treatment reduces chemotherapy-induced diarrhea and weight loss. Cancer Biol Ther. 2007 Sep;6(9):1449-54. doi: 10.4161/cbt.6.9.4622. Epub 2007 Jun 23. PMID 17881902
- [Background] Ciernikova S, Mego M, Semanova M, Wachsmannova L, Adamcikova Z, Stevurkova V, Drgona L, Zajac V. Probiotic Survey in Cancer Patients Treated in the Outpatient Department in a Comprehensive Cancer Center. Integr Cancer Ther. 2017 Jun;16(2):188-195. doi: 10.1177/1534735416643828. Epub 2016 May 5. PMID 27151581
- [Background] Ciorba MA, Hallemeier CL, Stenson WF, Parikh PJ. Probiotics to prevent gastrointestinal toxicity from cancer therapy: an interpretive review and call to action. Curr Opin Support Palliat Care. 2015 Jun;9(2):157-62. doi: 10.1097/SPC.0000000000000134. PMID 25872116
- [Background] Dai C, Zheng CQ, Meng FJ, Zhou Z, Sang LX, Jiang M. VSL#3 probiotics exerts the anti-inflammatory activity via PI3k/Akt and NF-kappaB pathway in rat model of DSS-induced colitis. Mol Cell Biochem. 2013 Feb;374(1-2):1-11. doi: 10.1007/s11010-012-1488-3. Epub 2012 Oct 23. PMID 23271629
- [Background] Dasari S, Kathera C, Janardhan A, Praveen Kumar A, Viswanath B. Surfacing role of probiotics in cancer prophylaxis and therapy: A systematic review. Clin Nutr. 2017 Dec;36(6):1465-1472. doi: 10.1016/j.clnu.2016.11.017. Epub 2016 Nov 24. PMID 27923508
- [Background] Escamilla J, Lane MA, Maitin V. Cell-free supernatants from probiotic Lactobacillus casei and Lactobacillus rhamnosus GG decrease colon cancer cell invasion in vitro. Nutr Cancer. 2012 Aug;64(6):871-8. doi: 10.1080/01635581.2012.700758. Epub 2012 Jul 25. PMID 22830611